## **Statistical Analysis Plan**

For

## A Pilot Study for the Evaluation of Minocycline as a Microglia Inhibitor in the Treatment of Branch Retinal Vein Occlusions

## NCT01468831

## Version 1.0 February 18, 2021

## Prepared by Megan Wall

| Original Author Signature: | |
|-----------------------------------|---------------------------|
| | Megan Wall, MS |
| Reviewer Signature: | |
| | Supriya Menezes, MS |
| Principal Investigator Signature: | |
| | Catherine Cukras, MD, PhD |

## TABLE OF CONTENTS

| LIS | ST OF ABBREVIATIONS | 3 |
|---|---|---|
| 1.0 | INTRODUCTION | |
| 1.1 | Branch Retinal Vein Occlusions (BRVO) | |
| 2.0 | DATA SOURCE | 5 |
| 3.0 | GENERAL REVIEW OF STUDY DESIGN | |
| 3.1 | Randomization, Masking and Unmasking | |
| 3.2 | Study Design | |
| 3.2.<br>3.2. | | |
| 3.2. | | |
| 3.3 | Study Objective | |
| 3.4 | Study Population | |
| 3.4. | .1 Inclusion Criteria | |
| 3.4. | | |
| 3.5 | | |
| 3.5. | | |
| 3.5. | · | |
| 3.5. | .3 Choice of Study Eye in Cases of Bilateral Eligibility Outcome Measures | |
| 3.6. | | |
| 3.6. | | |
| 3.6. | | |
| 4.0 | STATISTICAL CONSIDERATIONS | |
| 4.1 | Sample Size | |
| 4.2 | Analysis Population | |
| 4.3 | Descriptive Statistics | |
| 4.4 | Handling of Missing Values | |
| 4.5 | Handling Duplicate Assessments | |
| 4.6 | Software for Analyses | |
| 5.0 | PARTICIPANT DISPOSITION | |
| 6.0 | PARTICIPANT CHARACTERISTICS | |
| 6.1 | Participant Demographics | |
| 6.2 | Medical and Ophthalmic History | |
| 7.0 | PARTICIPANT COMPLIANCE | |
| 7.1 | Protocol Deviations and Unanticipated Problems | |
| 7.1.<br>7.2 | .1 IP Compliance Deviations | |
| 7.3 | Visit Schedule Deviations | |
| 8.0 | TREATMENT | |
| 9.0 | STOPPING THE STUDY | |
| 9.0<br>10.0 | PRIMARY OUTCOME ANALYSIS | |
| 10.0<br>11.0 | SECONDARY OUTCOMES ANALYSIS | |
| 11.0 | Number of Bevacizumab Injections | |
| 11.1 | Macular Sensitivity | |
| 11.3 | Best-Corrected Visual Acuity (BCVA) | |
| 11.4 | Optical Coherence Tomography (OCT) | |

## TABLE OF CONTENTS (CONTINUED)

| 11.5 | 1 - 6 | |
|---|---|---|
| 11.1 | Changes in Fluid Leakage | 25 |
| 12.0 | SAFETY ANALYSIS | |
| 12.1 | Adverse Events (AEs) | |
| 12.2 | | |
| | Doct Compated Visual Assitu (DCVA) | |
| 12.3<br>12.4 | Best-Corrected Visual Acuity (BCVA) Optical Coherence Tomography (OCT) | 26<br>26 |
| 12.4 | Intraocular Pressure (IOP) | |
| 12.6 | Thyroid Palpation Assessment and Review of Systems | |
| 12.7 | Laboratory Assessments | |
| 12.8 | Other Safety Outcomes | 27 |
| 13.0 | QUALITY ASSURANCE PLANS | 27 |
| 14.0 | REFERENCES | 28 |
| 15.0 | MOCK SHELLS | |
| 10.0 | NOCK CHELES | |
| | LIST OF TABLES | |
| Table 1 | : Participant Disposition | 29 |
| | Demographic Information by Site and Treatment Arm | |
| | : Medical and Ocular History | |
| | : Protocol Deviations and Unanticipated Problems | |
| | : Missed Study Procedures | |
| | : Missed and Out of Window Study Visits | |
| | : Analysis of Primary Outcome of Change in BCVA of the Study Eye from Baseline at Month | |
| , | | |
| Table 8 | 3: Analysis of Secondary Outcome of Number of Bevacizumab Injections by Participant from | |
| | Baseline to Month 12 and from Baseline to Month 24 | 34 |
| Table 9 | : Analysis of Secondary Outcome of Summary of Bevacizumab Injections by Treatment Arm | |
| | from Baseline to Month 12 and from Baseline to Month 24 | 34 |
| Table 1 | 0: Analysis of Secondary Outcome of Change in Macular Sensitivity as Measured by | |
| | Microperimetry from Baseline at Months 3, 6, 12, 18 and 24 | |
| Table 1 | 1: Analysis of Secondary Outcome of Change in BCVA of the Study Eye from Baseline at Mor | |
| Talala 1 | 24. | |
| rabie i | 2: Analysis of Secondary Outcome of Change in Central Retinal Thickness of the Study Eye from Baseline at Months 6, 12, 18 and 24 | |
| Tahla 1 | 3: Analysis of Secondary Outcome of Number of Participants Improving ≥ 1 logOCT Scale Ste | |
| 1 aute 1 | in the Study Eye at 12 and 24 Months Compared to Baseline | |
| Table 1 | 4: Analysis of Secondary Outcome of Change in Fluid Leakage in the Macula in the Study Eye | |
| 1 4010 1 | 12 and 24 Months Compared to Baseline | |
| Table 1 | 5: Summary of Adverse Events | |
| | 6: Summary of Adverse Events by System Organ Class (SOC) and Preferred Term (PT) | |
| | 7: Summary of Visual Acuity Over Time | |
| | 8: Summary of Central Retinal Thickness Over Time | |
| | 9: Summary of IOP Over Time | |
| 1 4010 1 | 2. 5 minutes 0. 101 0. 101 1. 111 0. 101 1. 111 0. 101 1. 111 0. 101 0. 101 | |

| Table 20: Results of Thyroid Palpation Assessment and Review of Systems Over Time | 39 |
|---|---|
| Table 21: Summary of Laboratory Assessments Over Time | 40 |
| LIST OF FIGURES | |
| Figure 1: Consort Diagram | 41 |
| Figure 2: Mean Best-Corrected Visual Acuity Over Time by Treatment Arm | 42 |
| Figure 3: Best-Corrected Visual Acuity Over Time by Participant | 43 |
| Figure 4: Mean Central Retinal Thickness Over Time by Treatment Arm | 43 |
| Figure 5: Central Retinal Thickness Over Time by Participant | 43 |
| LIST OF LISTINGS | |
| Listing 1: Demographic Information by Participant | 44 |
| Listing 2: IP Compliance | 44 |
| Listing A1. Visit Schedule Deviations Due to COVID-19 | 45 |

#### LIST OF ABBREVIATIONS

| Abbreviation | Definition |
|--------------|------------------------------------------------|
| AE | Adverse Event |
| APD | Afferent Pupillary Defect |
| BCVA | Best-Corrected Visual Acuity |
| BEH | Bristol Eye Hospital |
| BRC | Biomedical Research Centre |
| BRVO | Branch Retinal Vein Occlusion |
| BVOS | Branch Vein Occlusion Study |
| CFP | Color Fundus Photography |
| COVID-19 | Coronavirus Disease 2019 |
| CRVO | Central Retinal Vein Occlusion |
| CTCAE | Common Terminology Criteria for Adverse Events |
| CVA | Cerebral Vascular Event |
| DSMC | Data and Safety Monitoring Committee |
| ETDRS | Early Treatment Diabetic Retinopathy Study |
| FA | Fluorescein Angiography |
| FDA | Food and Drug Administration |
| HRVO | Hemi-Retinal Vein Occlusions |
| ICRRCC | Intramural Clinical Research Review Committee |
| IOP | Intraocular Pressure |
| IP | Investigational Product |
| IRB | Institutional Review Board |
| MedDRA | Medical Dictionary for Regulatory Activities |
| MI | Myocardial Infarction |
| NEI | National Eye Institute |
| OCT | Optical Coherence Tomography |
| PI | Principal Investigator |
| PRP | Panretinal Photocoagulation |
| PT | Preferred Term |
| RVO | Retinal Vein Occlusion |
| SAE | Serious Adverse Event |
| SD | Standard Deviation |
| SAP | Statistical Analysis Plan |
| SAS | Statistical Analysis Software |
| SOC | System Organ Class |
| VEGF | Vascular Endothelial Growth Factor |
| YAG | Yttrium Aluminum Garnet |

#### 1.0 Introduction

This statistical analysis plan (SAP) provides the proposed analyses for the MiBRVO protocol titled "A Pilot Study for the Evaluation of Minocycline as a Microglia Inhibitor in the Treatment of Branch Retinal Vein Occlusions". This document contains fifteen sections: (1) background of the study (2) data sources for analyses, (3) an overview of the study design, (4) statistical considerations, (5) participant disposition, (6) participant characteristics, (7) participant compliance, (8) treatment, (9) criteria for stopping the study, (10) statistical analysis for the primary outcome, (11) statistical abalysis for the secondary outcomes, (12) review of safety analyses, (13) quality assurance plans, (14) references, and (15) proposed data tables, figures and listings. This document is based on version 22.0 of the protocol dated December 10, 2019.

#### 1.1 Branch Retinal Vein Occlusions (BRVO)

Retinal vein occlusions (RVOs) are a significant source of vision loss, affecting mostly healthy people over 55 years of age. The common source of vision loss is the macular edema accompanying the retinal injury. The two main types of RVOs are branch retinal vein occlusions (BRVO) and central retinal vein occlusions (CRVO). Prevalence of BRVO, including hemi-retinal vein occlusions (HRVO), range between 0.6%-1.2% (1, 2). The fundamental cause of macular edema associated with RVOs is not completely understood, but it is increasingly clear that its pathophysiology extends beyond microvascular disease to involve immune mediators in the retina, such as microglia. Retinal microglia, derived from the monocytic lineage, are resident cells in the healthy retina that may be construed as representatives of the immune system in the immuneprivileged environment of the retina. There is accumulating evidence that retinal microglia are associated with inflammation in the retina in conditions such as diabetic retinopathy and the RVOs. Therefore, microglia represent a promising cellular target for forms of therapy that limit the deleterious inflammatory changes found in vein occlusions. Minocycline, a second-generation tetracycline with anti-inflammatory properties and high lipophilicity, appears to inhibit the activation of microglia as has been observed in animal studies and culture (3-6). Minocycline is used widely clinically and has been shown to be well tolerated when used as the FDA-approved doses proposed in this study. The objective of this study is to investigate the safety and potential efficacy of minocycline, a microglia inhibitor, in the treatment of BRVO.

#### 2.0 DATA SOURCE

Data received from the National Eye Institute (NEI) will be collected via their electronic data capture system (EMR), and uploaded on a daily basis to the Coordinating Center's database, Advantage EDC. Data received from the Bristol Eye Hospital (BEH) will be collected directly through Advantage EDC. Aligned OCT and microperimetry data collected for all participants will be provided directly to the Coordinating Center.

#### 3.0 GENERAL REVIEW OF STUDY DESIGN

## 3.1 Randomization, Masking and Unmasking

After the participant is determined eligible and has completed the informed consent process, the group will be assigned based on a predetermined randomization schedule developed by the Coordinating Center. Randomization will be stratified by site.

Randomization must occur on the same day as the initial administration of investigational product (IP) while the participant and the ophthalmologist are present and will not be permitted any time before. Participant eligibility must be confirmed before a participant is randomized. Participants will be randomized to one of two groups with equal probability for equal numbers of participants in each group: minocycline or placebo. Participants must continue to receive the same IP to which they were assigned for the duration of the study.

All clinic staff and participants will be masked to group assignments. Only designated pharmacy personnel, select individuals at the Emmes Company, LLC, and the NEI Data and Safety Monitoring Committee (DSMC) will have access to the group assignments.

Participants will be unmasked if deemed clinically necessary by the examining physician and if the study Principal Investigator (PI) and DSMC Chair are in agreement. In the case of a medical emergency, the examining or treating physician will have the final decision and unilateral right for unmasking. A request for unmasking, after approval by the PI and the DSMC Chair, will be made to Coordinating Center personnel, who will inform the PI and the DSMC Chair of the group assignment. Attempts should be made to maintain the masking of the investigators prior to the study-wide unmasking. Unmasking will be recorded on an adverse event (AE) form. All instances of unmasking must be reported to the ICRRC, the NIH IRB, and the DSMC. At the conclusion of the study, all investigators will be unmasked.

## 3.2 Study Design

For the NEI Site: The study duration will be 24 months. During this period, participants will be instructed to take the IP (either placebo or minocycline 100 mg capsule) twice daily. The primary outcome will be assessed at Month 12, and secondary outcomes will be assessed at 3, 6, 12, 18 and 24 months. Visits will occur at baseline, and then monthly or as clinically indicated. The study will require a minimum of 25 visits (baseline and Months 1-24). All appointments must be conducted within a window of ± seven days from the target day. The tests scheduled at each visit will be completed in one day. At each visit, the participant will undergo a review of systems and an assessment of safety variables. A complete ophthalmologic examination will be performed at each visit to measure outcome variables.

During each clinic visit, participants will have their visual acuity measured and will undergo optical coherence tomography (OCT) testing to measure retinal thickness.

For the Biomedical Research Centre (BRC) Sites: The study duration will be approximately 24 months. During this period, participants will be instructed to take the IP (either placebo or minocycline 100 mg capsule) twice daily. The primary outcome will be assessed at Month 12, and secondary outcomes will be assessed at 3, 6, 12, 18 and 24 months. Visits will occur at baseline, and then monthly or as clinically indicated. The study will require a minimum of 26 appointments (baseline and Months 1-24 and safety follow-up). All visits must be conducted within a window of  $\pm$  seven days from the target day, except the safety follow-up visit which must occur at least five days after the cessation of IP. The tests scheduled at each visit are expected to be completed in one day, with the exception of the baseline visit, Month 12 visit and Month 24 visit. If the baseline examinations cannot be performed in one clinic visit over one day, it is acceptable that the baseline examinations be completed at subsequent clinic visits, if scheduled within fourteen days of the first visit. If the Month 12 and Month 24 examinations cannot be performed in one clinic visit over one day, it is acceptable that the examinations be completed at subsequent clinic visits, if scheduled within seven days of the first visit. At each visit, the participant will undergo a review of systems and an assessment of safety variables. A complete ophthalmologic examination will be performed each visit (except for the safety follow-up visit) to measure outcome variables. If the baseline visit, Month 12 visit, or Month 24 visit are conducted over multiple days, bestcorrected visual acuity (BCVA), OCT and microperimetry testing must be conducted on the day

of the injection. If a participant or site is unable to complete microperimetry testing, the testing may be waived and the investigator will specify the reason the test could not be completed.

During each study visit, with the exception of the Month 24 visit and the safety follow-up visit at the BRC sites, IP will be dispensed to the participant unless the treatment is deemed to be "worsening" or to offer "no improvement" and the participant and the investigator decide to stop IP. An information sheet outlining instructions on taking the study medication and concomitant mediations will be distributed to participants and discussed in detail by study personnel. They will be asked to inform any physician who is prescribing new medications that they are currently taking minocycline. In addition, the participants will be asked to inform a study team member if a new medication is prescribed to them.

Participant compliance with IP will be prompted through ongoing encouragements and reminders during study visits and scheduled and unscheduled telephone contacts. Compliance will be assessed by pill counts conducted during study visits and the participant's pill diary.

Once identified, occurrences in which the computed compliance rate between study visits falls below 50% will be reported as a protocol deviation to the NIH IRB within two weeks using iRIS.

#### 3.2.1 Treatment Prior to Month 3

At baseline, the participant will receive an injection of 1.25 mg bevacizumab, an anti-vascular endothelial growth factor (VEGF) agent, and also start the randomized IP. At Months 1 and 2, the participant will again receive bevacizumab injections in the study eye and continue the randomized IP.

#### 3.2.2 Treatment Beginning at Month 3

Visual acuity and macular edema will be evaluated at study visits to determine further treatment. Starting at Month 3 and at every visit thereafter, the following scenarios will be considered. The participant will be re-injected with bevacizumab unless the participant meets the "improvement," "worsening," "new steady state" or "no improvement" criteria defined below.

Scenario 1: If the participant meets the "improvement" criteria, the participant will continue to take the IP, but the bevacizumab injection will be withheld at that visit.

Scenario 2: If the participant meets the "worsening" criteria, the participant will be offered any therapy available at the discretion of the treating investigator, including:

a. Focal Laser Treatment - If, based on fluorescein angiography, there is leakage into the fovea and insufficient focal laser treatment (i.e., extension of extra-foveal leakage beyond the lasered area), the participant may qualify for focal laser treatment. If the participant meets retreatment for focal laser, they can be retreated according to Branch Vein Occlusion Study (BVOS) guidelines if they have not been treated with focal laser in the past four months.

- b. Anti-VEGF Treatment.
- c. Intravitreal or Periocular Steroid Injections.

Scenario 3: If the participant does not meet the "improvement" or "worsening" criteria, but meets the "new steady state" criteria, the treating investigator physician will have the discretion to hold bevacizumab injections until the OCT changes (worsens) by > 25 microns from this "new steady state" level.

At the Month 12 visit and at every visit thereafter, Scenarios 1, 2 and 3 will be considered as well as the following scenario, which allows for a study physician to determine whether there has been "no improvement" in the participant's condition:

Scenario 4: If the participant meets the "no improvement" criteria or if the investigator's clinical impression is that there has been no improvement in the study eye, the participant will be offered therapy at the discretion of the treating investigator. The decision to re-inject the participant with bevacizumab (the anti-VEGF agent) will be made by the treating investigator after consulting with the participant. The decision to continue the IP will also be made by the treating investigator after consulting with the participant.

The "improvement," "worsening," "new steady state," and "no improvement" criteria are defined as follows:

- *Improvement*: Visual acuity in the study eye of ≥ 84-88 letters (20/20) OR OCT central subfield thickness <300 microns.
- Worsening: A decrease in visual acuity ≥ 15 or more letters in the study eye compared to baseline, AND an increase in OCT subfield thickness ≥ 1-step log unit compared to baseline for at least two consecutive visits.

• New steady state: Improvement and worsening criteria not met and central subfield thickness remains ≥ 300 microns on OCT, but thickness is stable and has not changed > 25 microns over the last three consecutive injections.

• *No improvement*: Improvement and worsening criteria are not met and visual acuity failed to increase by ≥ 10 letters in the study eye compared to baseline AND OCT central subfield thickness failed to decrease by ≥ 1-step log unit compared to baseline.

#### 3.2.3 Criteria for Stopping the Study

The DSMC may recommend temporarily suspending or closing enrollment, or stopping the study at any time due to safety concerns, demonstration of efficacy or lack of efficacy, or slow recruitment. Criteria for stopping the study include the following:

- A sufficiently large number of dropouts occurs as to make the trial likely to be uninformative;
- A participant experiences a drop in BCVA in the study eye of ≥ 30 letters from baseline attributed to the IP;
- A participant experiences a serious adverse event (SAE), drug reaction or complication, whether attributed to the IP or not, which has an impact on visual function or any other body system or precludes continuation of the IP. This would include the development of hypersensitization, allergic responses or other potentially serious drug reactions to medications required by the protocol.

Following premature IP discontinuation, not due to an AE, participants will continue to be followed as per the protocol.

#### 3.3 Study Objective

The objective of this study is to investigate the safety and potential efficacy of minocycline, a microglia inhibitor, in the treatment of BRVO.

#### 3.4 Study Population

A minimum of 10 and a maximum of 20 participants who meet the eligibility criteria may be enrolled from the NEI clinic and BEH sites, collectively. The recruitment totals are not fixed at either the NIH or BEH sites.

#### 3.4.1 Inclusion Criteria

To be eligible, the following inclusion criteria must be met, where applicable.

- 1. Participant is 18 years of age or older.
- 2. Participant must understand and sign the protocol's informed consent document.
- Female participants of childbearing potential must not be pregnant or breast-feeding and must be willing to undergo serum (BRC sites only) and urine pregnancy tests throughout the study.
- 4. <u>For the NEI Site</u>: Female participants of childbearing potential and male participants able to father children must have (or have a partner who has) had a hysterectomy or vasectomy, be completely abstinent from intercourse or must agree to practice two acceptable methods of contraception throughout the course of the study and for one week after study medication discontinuation (based on the half life of minocycline which is 11-22 hours). Acceptable methods of contraception include:
  - hormonal contraception (i.e., birth control pills\*, injected hormones, dermal patch or vaginal ring),
  - intrauterine device,
  - barrier methods (diaphragm, condom) with spermicide, or
  - surgical sterilization (hysterectomy or tubal ligation).

\*Oral birth control pills must be used with caution as minocycline decreases the effectiveness of some oral contraceptives. Participants already taking oral contraceptives may continue to use them, but must agree to use at least one other method of birth control while on study.

5. For the BRC Sites: Female participants of childbearing potential and male participants able to father children must have (or have a partner who has) had a hysterectomy or vasectomy or be completely abstinent from intercourse. Male participants or male partners (of female participants) who have not had a vasectomy or are not abstinent are required to use a condom with spermicide throughout the course of the study and for one week after study medication discontinuation (based on the half-life of minocycline which is 11-22 hours). Female participants of childbearing potential or female partners (of male participants) of childbearing potential must practice one of the below acceptable methods of contraception throughout the course of the study and for one week after study medication discontinuation:

- hormonal contraception (i.e., birth control pills\*, injected hormones, dermal patch or vaginal ring),
- intrauterine device,
- barrier methods (e.g., diaphragm) with spermicide, or
- surgical sterilization (hysterectomy or tubal ligation).

Abstinence is only acceptable when it is the participant's preferred and usual lifestyle choice. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception.

\*Oral birth control pills must be used with caution as minocycline decreases the effectiveness of some oral contraceptives. Participants already taking oral contraceptives may continue to use them but must agree to use at least one other method of birth control while on study.

It should be noted that two forms of contraception (as specified above) will be used by sexually active participants for the duration of the study and for one week after study medication discontinuation.

6. Participants must agree to notify the study investigator or coordinator if any of their doctors initiate a new medication during the course of the study.

7. Participant must have normal renal function and liver function or have mild abnormalities not above grade 1 as defined by the Common Terminology Criteria for Adverse Events v4.0 (CTCAE).

8. Participant has at least one eye that meets the study eye criteria listed in Section 3.4.

#### 3.4.2 Exclusion Criteria

A participant is not eligible if any of the following exclusion criteria are present.

- 1. Participant is in another investigational study and actively receiving IP for BRVO.
- 2. Participant is unable to comply with study procedures or follow-up visits.
- 3. Participant has a known hypersensitivity to sodium fluorescein dye.
- 4. Participant has a condition that, in the opinion of the investigator, would preclude participation in the study (e.g., unstable medical status including blood pressure and glycemic control).
- 5. Participant has a history of chronic renal failure requiring dialysis or kidney transplant.
- 6. Participant has a history of chronic hepatitis or liver failure.
- 7. Participant has an allergy or hypersensitivity to minocycline or any drug in the tetracycline family.
- 8. Participant is currently taking a tetracycline medication.
- 9. Participant is taking any medication that could adversely interact with minocycline such as methoxyflurane.
- 10. Participant has a blood pressure of > 180/110 (systolic above 180 **OR** diastolic above 110).
  - If blood pressure is brought below 180/110 by anti-hypertensive treatment, the participant can become eligible.
- 11. Participant is currently being treated with systemic anti-VEGF agents or systemic steroids.
- 12. Participant had a cerebral vascular event (CVA) or myocardial infarction (MI) within three months prior to study entry.
- 13. Participant has a history of thyroid cancer.

#### 3.5 Study Eye Eligibility Criteria

The participant must have at least one eye meeting all inclusion criteria and none of the exclusion criteria listed below.

## 3.5.1 Study Eye Inclusion Criteria

- 1. The study eye has a best-corrected Early Treatment Diabetic Retinopathy Study (ETDRS) visual acuity score between 78 and 34 letters (i.e., between 20/32 and 20/200).
- 2. The study eye shows evidence of definite retinal thickening due to a BRVO based on clinical examination involving the center of the macula that is not refractory to further therapy as based on the investigator's clinical judgment. BRVO is defined as an eye that had retinal hemorrhage or other biomicroscopic evidence of RVO (e.g., telangiectatic capillary bed) and a dilated (or previously dilated) venous system in one or two quadrants or less of the retina drained by the affected vein. HRVO is an RVO that involves two altitudinal quadrants. In this study, eyes with a HRVO will be considered a BRVO and are given the same treatment as BRVO eyes.
- 3. The study eye has retinal thickness in the central subfield on baseline OCT measurement > 350 microns, as measured by Zeiss Cirrus spectral domain OCT, or an equivalent retinal thickness on a similar OCT machine.
- 4. The study eye has media clarity and pupillary dilation sufficient for adequate fundus photographs. Furthermore, the participant must be able to cooperate during the procedure for accurate fundus photographs.

#### 3.5.2 Study Eye Exclusion Criteria

- 1. The study eye has macular edema considered to be due to a cause other than BRVO.
- 2. An eye should not be considered eligible if:
  - The macular edema is considered to be related to cataract extraction, or
  - Clinical examination and/or OCT suggest that vitreoretinal interface disease (e.g., a taut posterior hyaloid or epiretinal membrane) is the primary cause of the macular edema, or

• Clinical examination, medical history and/or fluorescein angiography suggest that diabetic retinopathy is the primary cause of the edema.

- 3. The study eye has a history of a recurrent RVO.
- 4. The study eye has a history of RVO present for > 18 months.
- 5. A brisk afferent pupillary defect (APD) is present in the study eye.
- 6. An ocular condition is present in the study eye such that, in the opinion of the investigator, visual acuity would not improve from resolution of macular edema (e.g., foveal atrophy, pigmentary changes, dense subfoveal hard exudates, laser scar at fovea, non-retinal condition).
- 7. An ocular condition (other than RVO) is present that, in the opinion of the investigator, might affect macular edema or alter visual acuity during the course of the study (e.g., uveitis or other ocular inflammatory disease, neovascular glaucoma, Irvine-Gass Syndrome, etc.).
- 8. A substantial cataract that, in the opinion of the investigator, is likely to be decreasing visual acuity by three lines or more (i.e., cataract would be reducing acuity to 20/40 or worse if eye was otherwise normal) is present in the study eye.
- 9. The study eye has had panretinal or sectoral scatter photocoagulation (PRP) within four months prior to study entry.
- 10. The study eye has had pars plana vitrectomy within six months prior to study entry.
- 11. The study eye has undergone major ocular surgery (including cataract extraction, scleral buckle, any intraocular surgery, etc.) within three months prior to study entry.
- 12. A yttrium aluminum garnet (YAG) capsulotomy has been performed on the study eye within two months prior to study entry.
- 13. The study eye has had treatment < three months prior to study entry of intravitreal or periocular steroid injections.
- 14. The study eye has had treatment < 28 days prior to study entry of intravitreal anti-VEGF agents.

## 3.5.3 Choice of Study Eye in Cases of Bilateral Eligibility

If both eyes of a participant meet the criteria described in Sections 3.5.1 and 3.5.2, the study eye will be determined at the investigator's discretion.

#### 3.6 Outcome Measures

#### 3.6.1 Primary Study Outcome

The primary outcome is the difference in mean change of BCVA, as measured in ETDRS letters, between the placebo and minocycline groups in the study eye at 12 months compared to baseline.

#### 3.6.2 Secondary Study Outcomes

Secondary outcomes include the difference between the minocycline and placebo groups in the:

- Number of bevacizumab injections from baseline to 12 months and from baseline to 24 months,
- Changes in mean macular sensitivity as measured by microperimetry at 3, 6, 12, 18 and 24 months compared to baseline,
- Mean change in the ETDRS BCVA in the study eye at 24 months compared to baseline,
- Changes in the retinal thickness in the study eye as measured by OCT at 6, 12, 18 and 24 months compared to baseline,
- Number of participants improving ≥ 1 logOCT scale step at 12 and 24 months compared to baseline,
- Changes in fluid leakage in the macular as demonstrated by fluorescein angiography at 12 and 24 months compared to baseline.

#### 3.6.3 Safety Outcomes

Safety outcomes will be the number and severity of systemic and ocular toxicities and AEs. The number of participants withdrawn from the IP due to vision loss or AEs and the number of participants deemed to have worsening disease will also contribute to the assessment of safety.

#### 4.0 STATISTICAL CONSIDERATIONS

## 4.1 Sample Size

No formal sample size has been calculated. The accrual ceiling for this study is 20 participants (10 per group) with a minimum of 10 participants (five per group). This number was selected to obtain at least five participants in each group reaching the final study visit in order to obtain preliminary data to potentially support a larger trial if possible if promising results are revealed.

## 4.2 Analysis Population

The following analysis populations will be considered for this study:

Enrolled population: Includes all participants enrolled in the study, regardless of compliance, follow-up or treatment received.

Safety population: Includes all participants who were exposed to IP, regardless of adherence to the protocol.

Primary outcome analysis population: Includes those participants who were exposed to IP and were followed up for at least 12 months.

#### 4.3 Descriptive Statistics

For continuous parameters, such as visual acuity, central retinal thickness as measured by OCT, and macular sensitivity as measured by microperimetry, descriptive statistics will include number of observations, mean, standard deviation, median, minimum and maximum. For categorical parameters, such as changes in fluid leakage as demonstrated by fluorescein angiography, frequency and percentage of participants will be summarized.

#### 4.4 Handling of Missing Values

If IP compliance cannot be determined for a participant due to missing capsule counts, IP compliance will be imputed by taking the median of all available capsule counts recorded at previous study visits.

If there are missing values for outcome data, then sensitivity analyses will be conducted as appropriate.

#### 4.5 Handling Duplicate Assessments

If participants completed assessments as both scheduled and supplementary visits, the assessments from the scheduled visit will be considered in the analysis and tabular summaries. However, if an assessment is completed only at supplementary visits, then the assessments from the most recent supplementary visit will be included in the analysis and tabular summaries. Results of all assessments, including those performed during supplementary visits, will be included in the listings.

#### 4.6 Software for Analyses

Statistical analyses will be performed using SAS version 9.4 or higher or R v3.6.1 or higher. All tables, listings and figures presented in the analysis will be created using either SAS v9.4 or Rv3.6.1 or higher.

#### 5.0 PARTICIPANT DISPOSITION

Overall participant disposition including the number and percentage of participants enrolled, completed 12 months of treatment, completed the study and discontinued the study early will be summarized. Reasons for study discontinuation will also be summarized (Table 1). The number and percentage of participants who withdraw from IP due to safety, including due to vision loss (manually identified based on investigator's comments for those participants with reason for withdrawal from IP indicated as "safety withdrawal") and AEs (reason for withdrawal from IP indicated as "safety withdrawal" for the occurrence of AEs assessed as being related to study IP that preclude further administration of IP) will be included. Further, the number and percentage of participants deemed to have worsening disease will be included. Worsening disease is defined as loss of 15 or more ETDRS letters of vision compared to baseline OR a  $\geq$  1-step increase in the logOCT scale. This table will be based on the enrolled population. Data will be presented by treatment and site.

Participant flow as outlined in Figure 1 will also be presented.

If a participant terminates from the study at Month 12 but completes the ophthalmic assessments as the Month 12 visit, they will be counted as having completed follow-up through Month 12. Similarly, if a participant discontinues IP or is deemed to have worsening disease at the Month 12 visit, the event will be considered to have occurred after Month 12.

#### 6.0 PARTICIPANT CHARACTERISTICS

These presentations will be based on the enrolled population.

## 6.1 Participant Demographics

Demographic characteristics including baseline age, sex, race and ethnicity. Demographic data will be summarized by treatment and site as outlined in Table 2 and listed in Listing 1. This table will be based on the enrolled population. The listing will include the registration date of participants as well as the eye that was selected to be the study eye and the treatment participants were randomized to.

#### 6.2 Medical and Ophthalmic History

The total number and percentage of participants with a history of medical and ocular conditions, medications, and ocular procedures will be summarized. History of ocular conditions and procedures will also be summarized by eye (study eye and fellow eye) and treatment (Table 3). Medical and ocular history will also be listed; the listing will include the date of diagnosis and/or time since diagnosis at baseline for select conditions and procedures.

Any findings from the physical examination at baseline will be included in a listing.

#### 7.0 PARTICIPANT COMPLIANCE

These presentations will be based on the enrolled population.

#### 7.1 Protocol Deviations and Unanticipated Problems

The total number of protocol deviations and unanticipated problems and the number and percentage of participants with deviations and unanticipated problems will be summarized. The number of events per participant and type (serious or not serious) and outcome of events will also be summarized (Table 4). Listings of participant specific and non-participant specific protocol deviations and unanticipated problems will be presented.

#### 7.1.1 IP Compliance Deviations

This listing will present the number of doses taken, the number of doses missed, the expected number of doses taken and the compliance rate for each participant (Listing 2). For each participant, the number of expected overall doses will be calculated as follows:

$$N_{Doses\ expected} = \left(Date_{Last\ study\ visit\ attended} - Date_{First\ date\ IP\ dispensed}\right) * 2$$

If participants took IP on the date they withdrew from the study or completed the study, the number of expected doses overall will be calculated as follows:

$$N_{Doses\ expected} = \left(Date_{Last\ study\ visit\ attended} - Date_{First\ date\ IP\ dispensed} + 1\right) * 2$$

If a participant disconinues IP between visits but continues in the study, the number of expected doses will be calculated as:

$$N_{Doses\ expected} = \left(Date_{Last\ date\ IP\ taken} - Date_{First\ date\ IP\ dispensed} + 1\right)*2$$

The sites will report the number of pills taken based on self-reported information as recorded in the pill diary. The number of doses taken and missed will be calculated for each participant as:

$$N_{Doses\ taken} = N_{Pills\ dispensed} - N_{Pills\ returned}$$

$$N_{Doses \ missed} = N_{Doses \ expected} - N_{Doses \ taken}$$

Negative values will indicate participants who took excess IP.

Compliance rates will be calculated as:

Compliance rate = 
$$(N_{Doses\ taken}/N_{Doses\ expected}) * 100$$

When IP compliance cannot be determined for a participant during any visit due to missing capsule counts, IP compliance will be imputed by taking the median of all available capsule counts recorded at previous study visits.

Participants with compliance rates less than 80% will be flagged.

#### 7.2 Study Procedure Deviations

This table will present the number of procedures not completed, the expected number of procedures completed, and the percentage of procedures missed by participant, procedure and collectively for all participants, cumulatively throughout the study (Table 5). Number of procedures not completed is defined when the site reports a missed procedure or when the protool monitors note a missed procedure at a site, and will be presented as a sum. Expected number of procedures completed is defined based on the study flowsheet included in the protocol, and will also be presented as a sum. Percentage of procedures missed will be calculated as follows:

$$(N_{procedures \, not \, completed}/N_{expected \, procedures \, completed}) * 100$$

#### 7.3 Visit Schedule Deviations

This table will present the number of expected visits, number of missed study visits, the percentage of missed study visits, the number of out of window visits, and the percentage of out of window visits for each individual participant and collectively for all participants, cumulatively throughout the study (Table 6). Number of expected, missed and out of window study visits will be calculated from the study flowsheet and will all be presented as sums. The percentage of missed study visits will be calculated as:

$$(N_{visits \, missed}/N_{expected \, visits}) * 100$$

Similarly, the percentage of out of window study visits will be calculated as:

Missed and out-of-window visits with the reason indicated as COVID-19 will also be presented by participant (Listing A1).

#### 8.0 TREATMENT

Information related to injections administered at each visit will be listed.

#### 9.0 STOPPING THE STUDY

If a participant meets one of the criteria for stopping the study listed in Section 3.2.3, a listing containing site, participant ID, date of last contact, visit number, reason for termination and comments related to termination will be constructed.

#### 10.0 PRIMARY OUTCOME ANALYSIS

The primary outcome is the difference in mean change of BCVA, as measured in ETDRS letters, between the placebo and minocycline groups in the study eye at 12 months compared to baseline. BCVA at baseline as well as change from baseline at Month 12 will be summarized for both treatment arms (Table 7). Interval estimates of mean change in BCVA will also be constructed as described below. The difference in mean change between the two groups at Month 12 will be calculated as the mean change from baseline at Month 12 for the Minocycline group minus the mean change from baseline at Month 12 for the Placebo group. Manifest refraction values for BCVA will be used when available.

Due to the small (N < 30) sample size, interval estimates for BCVA at baseline and Month 12 and change from baseline at Month 12 for each treatment group will be calculated as follows:

Confidence Interval = 
$$\bar{x} \pm t_{n-1,1-\alpha/2} * \sqrt{\frac{\sigma^2}{n}}$$

Where:

 $\bar{x}$  is the mean.

t  $_{n-1, 1-\alpha/2}$  is the t-value with n-1 degrees of freedom at a confidence level of  $\alpha$ .

n is the number of observations.

 $\sigma$  is the standard deviation.

Additionally, due to the small (N < 30) sample size, interval estimates for the mean difference in BCVA at baseline and Month 12 between the two groups as well as the difference in the mean change in BCVA from baseline at Month 12 bewteen the two groups will be calculated as follows:

Confidence Interval = 
$$(\overline{x_1} - \overline{x_2}) \pm t_{d,1-\alpha/2} * \sqrt{\sigma_{T1-T2}^2}$$

Where:

 $\overline{x_1}$  and  $\overline{x_2}$  are the means for the Minocycline and Placebo groups, respectively.

 $t_{d, 1-\alpha/2}$  is the t-value with d degrees of freedom at a confidence level of  $\alpha$ . d will be determined using the below equation.

 $\sigma_{T1-T2}$  is the standard deviation of the difference between the means of the Minocycline and Placebo groups and will be calculated using the below equation.

The degrees of freedom, d, for the t-value used to calculate the confidence interval of the difference between the two groups will be determined as follows:

$$d = \frac{\left(\frac{\sigma_1^2}{n_1} + \frac{\sigma_2^2}{n_2}\right)^2}{\frac{1}{n_1 - 1} \left(\frac{\sigma_1^2}{n_1}\right)^2 + \frac{1}{n_2 - 1} \left(\frac{\sigma_2^2}{n_2}\right)^2}$$

Where:

 $\sigma_1$  and  $\sigma_2$  are the standard deviations for the Minocycline and Placebo groups, respectively.  $n_1$  and  $n_2$  are the number of observations of the Minocycline and Placebo groups, respectively.

The standard deviation of the difference between the means of the Minocycline and Placebo groups will be calculated as follows:

$$\sigma_{T1-T2} = \sqrt{\frac{\sigma_1^2}{n_1} + \frac{\sigma_2^2}{n_2}}$$

Where:

 $\sigma_1$  and  $\sigma_2$  are the standard deviations for the Minocycline and Placebo groups, respectively.  $n_1$  and  $n_2$  are the number of observations of the Minocycline and Placebo groups, respectively.

This analysis will be based on the primary outcome analysis population.

Additional presentations stratified by site will be constructed as appropriate.

Exploratory statistical analyses will be conducted as appropriate.

Participants who were exposed to recent (< three months) systemic steroid or systemic anti-VEGF prior to enrolling will be analyzed separately as appropriate to assess for any possible confounding effects for treatment benefit.

#### 11.0 SECONDARY OUTCOMES ANALYSIS

These analyses will be based on the safety population who completed the respective visits.

Additional presentation stratified by site will be constructed as appropriate.

Exploratory statistical analyses will be conducted as appropriate.

Participants who were exposed to recent (< three months) systemic steroid or systemic anti-VEGF prior to enrolling will be analyzed separately as appropriate to assess for any possible confounding effects for treatment benefit.

#### 11.1 Number of Bevacizumab Injections

The number of bevacizumab injections from baseline to 12 months and from baseline to 24 months will be tabulated by participant (Table 8). Additionally, the average number of injections between baseline and Months 12 and 24 will be calculated for each treatment arm, and the difference in the number of injections between the two groups will be presented (Table 9). The difference in the number of injections between the two groups will be calculated as the number of injections in the Minocycline group minus the number of injections in the Placebo group.

#### 11.2 Macular Sensitivity

Mean change in macular sensitivity in the study eye, as measured by microperimetry, from baseline at Months 3, 6, 12, 18 and 24 will be summarized by treatment arm, and interval estimates will be constructed (Table 10). The difference in mean macular sensitivity between the two groups will also be presented. Interval estimates will be calculated using the method described in Section 10.0. The mean difference in macular sensitivity between the two groups at a visit will be calculated as the mean change from baseline in the Minocycline group minus the mean change from baseline in the Placebo group.

#### 11.3 Best-Corrected Visual Acuity (BCVA)

The mean change in ETDRS BCVA of the study eye at 24 months compared to baseline will be analyzed similar to the primary outcome detailed in Section 10.0 (Table 11). Manifest refraction values for BCVA will be used when available.

## 11.4 Optical Coherence Tomography (OCT)

The changes in retinal thickness in the study eye, as measured by aligned OCT, at 6, 12, 18 and 24 months compared to baseline will be summarized by treatment arm, and interval estimates will be constructed (Table 12). The difference in retinal thickness between the two groups will also be presented. Interval estimates will be calculated using the method described in Section 10.0. The difference in retinal thickness between the two groups at a visit will be calculated as the mean change from baseline in the Minocycline group minus the mean change from baseline in the Placebo group.

#### 11.5 Improvement of ≥ 1 logOCT Scale Step

The number of participants improving  $\geq 1 \log OCT$  scale step at 12 and 24 months compared to baseline in the study eye will be presented by treatment arm (Table 13). The difference in the number of participants improving  $\geq 1 \log OCT$  scale step from baseline will be calculated as the number of participants improving in the Minocycline group minus the number of participants improving in Placebo group and will use aligned OCT.

Improvement of  $\geq 1$  logOCT scale step is defined as a decrease of  $\geq 1$ -step on the logOCT scale, where:

$$LogScore = 10 * log_{10}(thickness/300)$$

 $Step\ change\ on\ log OCT\ scale = Log Score_{Follow\ up} - Log Score_{Baseline}$ 

A decrease in one-step is considered clinically significant (7). A one-step decrease is equivalent to at least a 20% improvement of central macular thickness and represents greater than twice the variability of retinal thickness measurements (approximately 25-30 microns). The table below presents examples of OCT measurements with their corresponding LogScore.

**OCT and Corresponding LogScores (7)** 

| LogScore | OCT (µm) |
|----------|----------|
| 0 | 300 |
| 0.5 | 337 |
| 1 | 378 |
| 1.5 | 424 |
| 2 | 475 |
| 2.5 | 533 |
| 3 | 599 |
| 3.5 | 672 |
| 4 | 754 |
| 4.5 | 846 |
| 5 | 949 |
| 5.5 | 1064 |
| 6 | 1194 |
| 6.5 | 1340 |

#### 11.1 Changes in Fluid Leakage

Changes in the fluid leakage in the macula of the study eye, as demonstrated by fluorescein angiography, at 12 and 24 months compared to baseline will be summarized by treatment arm (Table 14). The difference in changes in fluid leakage between the two groups will also be presented as the change in fluid leakage in the Minocycline group minus the change in fluid leakage in Placebo group.

#### 12.0 SAFETY ANALYSIS

These analyses will be based on the safety population, unless otherwise specified. All relevant information will be listed; data for all enrolled participants will be included in the listings. Relevant data may be plotted against time.

Additional presentations stratified by site will be constructed as appropriate.

#### 12.1 Adverse Events (AEs)

All AEs reported will be summarized by treatment arm and overall. Total number and percentage of participants with AEs will be presented by severity, ocular specification, outcome, and relation to IP (Table 15). AEs will also be summarized by system organ class (SOC) and preferred term (PT) (Table 16). If sufficient data is present, summaries similar to Table 15 and Table 16 will be generated for all serious adverse events (SAEs), and summaries similar to Table 16 will be presented for natural progression of the disease.

All AEs and events corresponding to natural progressions of the disease will be listed.

# 12.2 Withdrawal from IP Due to Vision Loss and Adverse Events and Participants with Worsening Disease

Participants who discontinue IP due to vision loss and adverse events will be summarized in Table 1. Participants who are deemed to have worsening disease in the study or fellow eye at any point during follow-up will also be presented in Table 1. Worsening disease is defined as a loss of 15 or more ETDRS letters of vision compared to baseline OR a 1-step increase in the logOCT scale.

#### 12.3 Best-Corrected Visual Acuity (BCVA)

Visual acuity will be collected at baseline and all follow-up visits for both eyes. Total letters read at each visit and change from baseline at each follow-up visit will be presented overall and by treatment arm for both the study and fellow eyes in Table 17. The number and percentage of participants with  $\geq 10$  letter change at each visit will also be included. Manifest refraction values for BCVA will be used when available.

Mean BCVA will be plotted over time for the minocycline and placebo treatment arms for both the study and fellow eyes (Figure 2). Individual BCVA will also be plotted over time for both eyes (Figure 3).

## 12.4 Optical Coherence Tomography (OCT)

Central retinal thickness, as measured by OCT, is assessed at all visits for both eyes. Central retinal thickness and change from baseline at each follow-up visit will be presented overall and by treatment arm for the study and fellow eyes in Table 18.

Mean central retinal thickness will be plotted over time for the minocycline and placebo treatment arms for both the study and fellow eyes (Figure 4). Individual central retinal thickness will also be plotted over time for both eyes (Figure 5).

#### 12.5 Intraocular Pressure (IOP)

Intraocular pressure (IOP) is assessed at all visits for both eyes. IOP measurements at each visit and change from baseline at each follow-up visit will be summarized using descriptive statistics and will be presented overall and by treatment arm for both the study and fellow eyes (Table 19).

#### 12.6 Thyroid Palpation Assessment and Review of Systems

A thyroid palpation assessment and a review of systems is completed at every visit. The number and percentage of participants with clinically significant thyroid palpation findings will be summarized overall and by treatment arm (Table 20). The number of percentage of participants who experienced dizziness, sun sensitivity, or diarrhea between visits will also be summarized in Table 20.

#### 12.7 Laboratory Assessments

An acute care panel, hepatic panel and thyroid function testing will be performed at baseline, Month 2 and every four months thereafter (Months 6, 10, 14, 18 and 22), as well as the final visit at Month 24. Frequency and percentage of participants reporting laboratory abnormalities at baseline will be summarized with shift from baseline to each follow-up visit (Table 21).

#### 12.8 Other Safety Outcomes

Exploratory analyses and/or descriptive summary statistics of color fundus photography (CFP), fluorescein angiogram (FA), microperimetry and other assessments will be performed as appropriate.

#### 13.0 QUALITY ASSURANCE PLANS

To ensure accurate, reliable study results, two statisticians will separately analyze and compare the primary study outcome. All SAS or R code used to generate primary and secondary outcomes will undergo a code validation by an independent statistician or SAS programmer. Documentation related to code validation audits will be maintained on file at the Coordinating Center.

#### 14.0 REFERENCES

 Mitchell P, Smith W, Chang A. Prevalence and associations of retinal vein occlusion in Australia. The Blue Mountains Eye Study. Archives of ophthalmology 1996; 114(10): 1243-1247

- 2. Klein R, Klein BE, Moss SE, Meuer SM. The epidemiology of retinal vein occlusion: the Beaver Dam Eye Study. Transactions of the American Ophthalmological Society 2000; 98: 133-141; discussion 141-133.
- 3. Zemke D, Majid A. The potential of minocycline for neuroprotection in human neurologic disease. Clin Neuropharmacol 2004; 27(6): 293-298.
- 4. Tikka T, Fiebich BL, Goldsteins G, Keinanen R, Koistinaho J. Minocycline, a tetracycline derivative, is neuroprotective against excitotoxicity by inhibiting activation and proliferation of microglia. J Neurosci 2001; 21(8): 2580-2588.
- 5. Bosco A, Inman DM, Steele MR et al. Reduced retina microglial activation and improved optic nerve integrity with minocycline treatment in the DBA/2J mouse model of glaucoma. Investigative ophthalmology & visual science 2008; 49(4): 1437-1446.
- 6. Yang LP, Zhu XA, Tso MO. A possible mechanism of microglia-photoreceptor crosstalk. Molecular vision 2007; 13: 2048-2057.
- 7. Ferris FL 3rd, Miller KM, Glassman AR, Beck RW; Diabetic Retinopathy Clinical Research Network. A proposed method of logarithmic transformation of optical coherence tomography data for use in clinical research. Ophthalmology. 2010 Aug;117(8): 1512-6.

#### 15.0 MOCK SHELLS

#### **TABLES**

**Table 1: Participant Disposition** 

| | ВЕН | | | NEI | | | Total | | |
|---|---|---|---|---|---|---|---|---|---|
| | Minocycline | Placebo | Total | Minocycline | Placebo | Total | Minocycline | Placebo | Total |
| Disposition | $(N=X)^1$ | $(N=X)^1$ | $(N=X)^1$ | $(N=X)^1$ | $(N=X)^1$ | $(N=X)^1$ | $(N=X)^1$ | $(N=X)^{1}$ | $(N=X)^1$ |
| Enrolled | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) |
| Completed Follow-up Through Month 12 | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) |
| <b>Completed Study</b> | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) |
| Completed Follow-up | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) |
| Terminated per protocol | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) |
| Discontinued IP Early | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) |
| Prior to Month 12 | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) |
| After Month 12 | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) |
| Reason | | | | | | | | | |
| Participant non-compliance | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) |
| Safety Withdrawal | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) |
| Vision loss <sup>2</sup> | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) |
| $AEs^3$ | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) |
| Other | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) |
| Discontinued Study Early | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) |
| Prior to Month 12 | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) |
| After Month 12 | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) |
| Reason | | | | | | | | | |
| AE/intercurrent illness | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) |
| Death | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) |
| Requested termination | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) |
| Other | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) |
| Deemed to Have Worsening Disease <sup>4,5</sup> | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) |
| Prior to Month 12 <sup>5</sup> | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) |
| Study Eye | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) |
| Fellow Eye | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) |
| After Month 12 <sup>5</sup> | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) |
| Study Eye | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) |
| Fellow Eye | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) |

<sup>1</sup> Column header counts and denominators are the number of participants in the enrolled population in each treatment arm and overall. Percentages are rounded to the nearest whole number.

<sup>&</sup>lt;sup>2</sup> Manually identified based on investigator's comments for those participants with reason for withdrawal from IP as "safety withdrawal".

<sup>&</sup>lt;sup>3</sup> Participants with reason for withdrawal from IP indicated as "safety withdrawal" for the occurrence of AEs assessed as being related to the study IP that preclude further administration of IP.

<sup>&</sup>lt;sup>4</sup> Worsening disease is defined as a loss of 15 or more ETDRS letters of vision compared to baseline OR a 1-step increase in the logOCT scale.

<sup>&</sup>lt;sup>5</sup> If a participant experienced worsening disease in both the study and fellow eyes, the participant will only be counted once.

**Table 2: Demographic Information by Site and Treatment Arm** 

| | ВЕН | | | | NEI | | | Total | |
|---|---|---|---|---|---|---|---|---|---|
| | Minocycline | Placebo | Total | Minocycline | Placebo | Total | Minocycline | Placebo | Total |
| <b>Demographic Characteristics</b> | $(N=X)^1$ | $(N=X)^1$ | $(N=X)^1$ | $(N=X)^1$ | $(N=X)^1$ | $(N=X)^1$ | $(N=X)^1$ | $(N=X)^1$ | $(N=X)^1$ |
| Gender N (%) | , , | , | | , , , | , | • | , , , | , | , |
| Female | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) |
| Male | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) |
| Age Category (years) at Baseline N (%) | | | | | | | | | |
| 56-60 | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) |
| 61-65 | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) |
| 66-70 | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) |
| 71-75 | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) |
| 76-80 | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) |
| 81-85 | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) |
| Age (years) at Baseline | , , | ` , | . , | , , | , , | ` , | ` ' | , , | ` , |
| N | X | X | X | X | X | X | X | X | X |
| Mean (SD) | x.x(x.x) | x.x(x.x) | x.x(x.x) | x.x(x.x) | x.x(x.x) | x.x(x.x) | x.x(x.x) | x.x(x.x) | x.x(x.x) |
| Median | X | X | X | X | X | X | X | X | X |
| Range (Min, Max) | (x, x) | (x, x) | (x, x) | (x, x) | (x, x) | (x, x) | (x, x) | (x, x) | (x, x) |
| Ethnicity N (%) | , , , | | | , , , | | | | | |
| Hispanic or Latino | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) |
| Not Hispanic or Latino | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) |
| Unknown | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) |
| Race N (%) | , , | ` , | . , | , , | , , | ` , | ` ' | , , | ` , |
| American Indian or Alaskan Native | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) |
| Asian | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) |
| Black | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) |
| Hawaiian or Pacific Islander | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) |
| White | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) |
| Multiple Race | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) |
| Unknown | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) |

<sup>&</sup>lt;sup>1</sup> Column header counts and denominators are the number of participants in the enrolled population in each treatment arm and overall. Percentages are rounded to the nearest whole number.

**Table 3: Medical and Ocular History** 

| | | Minocycline | | | Placebo | | Total | | |
|---|---|---|---|---|---|---|---|---|---|
| Conditions/Procedures | Study Eye<br>(N=X) <sup>1</sup> | Fellow Eye<br>(N=X) <sup>1</sup> | Total (N=X) <sup>1,2</sup> | Study Eye<br>(N=X) <sup>1</sup> | Fellow Eye (N=X) <sup>1</sup> | Total (N=X) <sup>1,2</sup> | Study Eye<br>(N=X) <sup>1</sup> | Fellow Eye (N=X) <sup>1</sup> | Total (N=X) <sup>1,2</sup> |
| Any Medical Condition | , | , | x (x%) | , | , , | x (x%) | , | , , | x (x%) |
| Renal disease | | | , | | | , | | | , , |
| Yes | | | x (x%) | | | x (x%) | | | x (x%) |
| No | | | x (x%) | | | x (x%) | | | x (x%) |
| Hepatitis | | | | | | | | | |
| Yes | | | x (x%) | | | x (x%) | | | x (x%) |
| No | | | x (x%) | | | x (x%) | | | x (x%) |
| Any Medication History Systemic anti-VEGF | | | x (x%) | | | x (x%) | | | x (x%) |
| Yes | | | x (x%) | | | x (x%) | | | x (x%) |
| No | | | x (x%) | | | x (x%) | | | x (x%) |
| Systemic steroid | | | (, -) | | | (, -) | | | (, -) |
| Yes | | | x (x%) | | | x (x%) | | | x (x%) |
| No | | | x (x%) | | | x (x%) | | | x (x%) |
| Any Ocular Condition Recurrent RVO | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) |
| Yes | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) |
| No | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) |
| RVO present > 18 months | ` ′ | , , | | | | • | ` | | , , , |
| Yes | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) |
| No | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) |
| Any Ocular Procedure Intravitreal steroid injection | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) |
| Yes | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) |
| No | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) |
| Cataract surgery | ` / | , | , | ` / | , | ` / | ` / | , | , |
| Yes | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) |
| No | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) |
| ••• | ` / | · / | ` / | . / | ` / | ` / | ` / | ` / | ` / |

<sup>&</sup>lt;sup>1</sup> Column header counts and denominators are the number of participants in the enrolled population in each treatment arm and overall. Percentages are rounded to the nearest whole number. <sup>2</sup> If a participant reported an ocular condition or procedure in both eyes, the participant will only be counted only once.

**Table 4: Protocol Deviations and Unanticipated Problems** 

| | Partic | ipant-Specific | Non-Participant Specific | Total |
|---|---|---|---|---|
| | N | Sumber of Participants | | |
| | Number of | with Events | Number of | Number of |
| | <b>Events</b> | $(N=X)^1$ | Events | <b>Events</b> |
| All Events | X | x (x%) | х | X |
| Protocol Deviations | X | x (x%) | X | X |
| Unanticipated Problems | X | $x(x^{0/0})$ | X | X |
| Number of Events per Participant | | | | |
| Mean (SD) | x.x(x.x) | | | |
| Median | X | | | |
| Range (Min, Max) | x, x | | | |
| Туре | | | | |
| Serious | X | x (x%) | X | X |
| Not serious | X | x(x%) | X | X |
| Outcome | | | | |
| Participant follow-up continues | X | x (x%) | X | X |
| Participant follow-up terminated | X | x(x%) | X | X |
| | X | x(x%) | X | X |

<sup>&</sup>lt;sup>1</sup> Column header count and denominators are the number of participants in the enrolled population. Percentages are rounded to the nearest whole number.

**Table 5: Missed Study Procedures** 

| Category | Site | Participant ID/<br>Procedure | Number of<br>Expected<br>Procedures | Number of<br>Missed<br>Procedures | Percentage of<br>Missed<br>Procedures |
|---|---|---|---|---|---|
| Participant | XXX | 001 | XX | XX | X.X |
| | XXX | 002 | XX | XX | X.X |
| | XXX | 003 | XX | XX | X.X |
| | | ••• | XX | XX | X.X |
| | | | XX | XX | X.X |
| Procedure | | Acute Care Panel | xx | XX | X.X |
| | | Adverse Event<br>Assessment | xx | xx | X.X |
| | | BCVA (ETDRS) | XX | XX | X.X |
| | | ••• | XX | XX | X.X |
| | | | XX | XX | X.X |
| Total | | | XX | XX | <b>x.</b> x |

**Table 6: Missed and Out of Window Study Visits** 

| Site | Participant<br>ID | Number of<br>Expected Visits | Number of<br>Missed Visits | Percentage of<br>Missed Visits | Number of Out<br>of Window<br>Visits | Percentage of<br>Out of Window<br>Visits | Visits Missed or<br>Out of Window |
|---|---|---|---|---|---|---|---|
| XXX | 001 | XX | XX | X.X | XX | X.X | XXX |
| XXX | 002 | XX | XX | X.X | XX | X.X | |
| ••• | ••• | XX | XX | X.X | XX | X.X | |
| Total | | XX | XX | X.X | XX | X.X | |

Table 7: Analysis of Primary Outcome of Change in BCVA of the Study Eye from Baseline at Month 12

| | Minoc | cycline | Plac | cebo | Differ | Difference <sup>1</sup> |
|---|---|---|---|---|---|---|
| | BCVA | Δ | BCVA | Δ | BCVA | Δ |
| Visit | (letters read) | (letters read) | (letters read) | (letters read) | (letters read) | (letters read) |
| Baseline | | | | | | |
| N | X | | X | | | |
| Mean (SD) | x (x) | | x (x) | | x (x) | |
| 95% Confidence Interval | (x, x) | | (x, x) | | (x, x) | |
| Month 12 | | | | | | |
| N | X | X | X | X | | |
| Mean (SD) | x(x) | x (x) | x (x) | x (x) | x (x) | x (x) |
| 95% Confidence Interval | (x, x) | (x, x) | (x, x) | (x, x) | (x, x) | (x.x, x.x) |

 $<sup>\</sup>Delta$  indicates change from baseline.

<sup>&</sup>lt;sup>1</sup> Difference is defined as the Minocycline – Placebo treatment arms. Negative values indicate that participants in the Placebo group experienced a higher visual acuity or a more positive change from baseline at Month 12.

Table 8: Analysis of Secondary Outcome of Number of Bevacizumab Injections by Participant from Baseline to Month 12 and from Baseline to Month 24

| Site | Participant ID | Treatment Arm | Visit Period | Number of Bevacizumab Injections |
|---|---|---|---|---|
| XXX | 001 | Minocycline/Placebo | Baseline to Month 12 | XX |
| | | • | Baseline to Month 24 | XX |
| xxx | 002 | Minocycline/Placebo | Baseline to Month 12 | XX |
| | | | Baseline to Month 24 | XX |
| | ••• | | | |

Table 9: Analysis of Secondary Outcome of Summary of Bevacizumab Injections by Treatment Arm from Baseline to Month
12 and from Baseline to Month 24

| | Minocycline | Placebo | |
|----------------------|-------------|-----------|-------------------------|
| Visit Period | $(N=X)^1$ | $(N=X)^1$ | Difference <sup>2</sup> |
| Baseline to Month 12 | | | |
| Number of Injections | XX | XX | XX |
| Mean | X.X | X.X | X.X |
| Baseline to Month 24 | | | |
| Number of Injections | XX | XX | XX |
| Mean | X.X | X.X | X.X |

<sup>&</sup>lt;sup>1</sup> Column header counts are the number of participants in the safety population in each treatment arm and overall.

<sup>&</sup>lt;sup>2</sup> Difference is defined as the Minocycline – Placebo treatment arms. Negative values indicate that participants in the Placebo group received more injections during the respective visit period.

# Table 10: Analysis of Secondary Outcome of Change in Macular Sensitivity as Measured by Microperimetry from Baseline at Months 3, 6, 12, 18 and 24

This table will be similar to Table 7.

# Table 11: Analysis of Secondary Outcome of Change in BCVA of the Study Eye from Baseline at Month 24

This table will be similar to Table 7.

# Table 12: Analysis of Secondary Outcome of Change in Central Retinal Thickness of the Study Eye from Baseline at Months 6, 12, 18 and 24

This table will be similar to Table 7.

Table 13: Analysis of Secondary Outcome of Number of Participants Improving ≥ 1 logOCT Scale Step in the Study Eye at 12 and 24 Months Compared to Baseline

| Visit | Minocycline<br>N (%) <sup>1</sup> | Placebo<br>N (%) <sup>1</sup> | Difference <sup>2</sup> |
|---|---|---|---|
| Month 12 | x (x%) | x (x%) | X |
| Month 24 | x (x%) | x(x%) | X |

<sup>&</sup>lt;sup>1</sup> Denominators are the number of participants in the safety population in each treatment arm and overall with data at the given visit. Percentages are rounded to the nearest whole number.

Table 14: Analysis of Secondary Outcome of Change in Fluid Leakage in the Macula in the Study Eye at 12 and 24 Months Compared to Baseline

| Visit | Minocycline | Placebo | Difference <sup>2</sup> |
|---|---|---|---|
| Visit | N (%) <sup>1</sup> | N (%) <sup>1</sup> | Difference |
| Month 12 | | | |
| Increase | x (x%) | x (x%) | X |
| Decrease | x(x%) | x(x%) | X |
| No Change | x (x%) | x (x%) | X |
| Month 24 | | | |
| Increase | x (x%) | x (x%) | X |
| Decrease | x (x%) | x (x%) | X |
| No Change | x(x%) | x(x%) | X |

<sup>&</sup>lt;sup>1</sup> Denominators are the number of participants in the safety population in each treatment arm and overall with data at the given visit. Percentages are rounded to the nearest whole number.

<sup>&</sup>lt;sup>2</sup> Difference is defined as Minocycline – Placebo treatment arms. Negative values indicate that more participants in the Placebo group improved by  $\geq 1$  logOCT scale step at the respective visit compared to baseline.

<sup>&</sup>lt;sup>2</sup> Difference is defined as Minocycline – Placebo treatment arms. Negative values indicate that more participants in the Placebo group experienced a certain change in fluid leakage at the respective visit compared to baseline.

**Table 15: Summary of Adverse Events** 

| | Minoc | ycline | Plac | ebo | To | tal |
|---|---|---|---|---|---|---|
| | Participants with Events N (%) <sup>1</sup> | Number of<br>Events<br>N | Participants with Events N (%) <sup>1</sup> | Number of<br>Events<br>N | Participants with Events N (%) <sup>1</sup> | Number of<br>Events<br>N |
| All AEs | x (x%) | X | x (x%) | X | x (x%) | X |
| Serious Adverse Events | x (x%) | X | x (x%) | X | x (x%) | X |
| Severity | | | | | | |
| Mild | x (x%) | X | x (x%) | X | x (x%) | X |
| Moderate | x (x%) | X | x (x%) | X | x (x%) | X |
| Severe | x (x%) | X | x (x%) | X | x (x%) | X |
| Life-threatening | x (x%) | X | x (x%) | X | x (x%) | X |
| Death | x (x%) | X | x (x%) | X | x (x%) | X |
| Eye | | | | | | |
| Non-ocular | x (x%) | X | x (x%) | X | x (x%) | X |
| Study eye | x (x%) | X | x (x%) | X | x (x%) | X |
| Fellow eye | x (x%) | X | x (x%) | X | x (x%) | X |
| Outcome | | | | | | |
| Resolved | x (x%) | X | x (x%) | X | x (x%) | X |
| Resolved with sequalae | x (x%) | X | x (x%) | X | x (x%) | X |
| Death | x (x%) | X | x (x%) | X | x (x%) | X |
| Resolved by convention | x (x%) | X | x (x%) | X | x (x%) | X |
| Relation to IP | | | | | | |
| Yes | x (x%) | X | x (x%) | X | x (x%) | X |
| No | x (x%) | X | x (x%) | X | x (x%) | X |

<sup>&</sup>lt;sup>1</sup> Denominators are the number of participants in the safety population in each treatment arm and overall. Percentages are rounded to the nearest whole number.

Table 16: Summary of Adverse Events by System Organ Class (SOC) and Preferred Term (PT)

| Minoc | ycline | Plac | ebo | Total | |
|---|---|---|---|---|---|
| Participants with Events N (%) <sup>1</sup> | Number of<br>Events<br>N | Participants<br>with Events<br>N (%) <sup>1</sup> | Number of<br>Events<br>N | Participants<br>with Events<br>N (%) <sup>1</sup> | Number of<br>Events<br>N |
| x (x%) | X | x (x%) | X | x (x%) | X |
| x (x%) | X | x (x%) | X | x(x%) | X |
| x (x%) | X | x(x%) | X | x(x%) | X |
| x (x%) | X | x (x%) | X | x(x%) | X |
| x (x%) | X | x (x%) | X | x (x%) | X |
| ` / | X | ` / | X | ` ' | X |
| - | Participants with Events N (%)¹ x (x%) x (x%) x (x%) x (x%) | with Events Events N (%)¹ N x (x%) x x (x%) x | Participants with Events Number of Events Participants with Events N (%)¹ N N (%)¹ x (x%) x x (x%) x (x%) x x (x%) x (x%) x x (x%) x (x%) x x (x%) x (x%) x x (x%) x (x%) x x (x%) | $ \begin{array}{c ccccccccccccccccccccccccccccccccccc$ | $ \begin{array}{c ccccccccccccccccccccccccccccccccccc$ |

<sup>1</sup> Denominators are the number of participants in the safety population in each treatment arm and overall. Percentages are rounded to the nearest whole number.

**Table 17: Summary of Visual Acuity Over Time** 

| | | Minoc | cycline | | | Plac | cebo | | | To | tal | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | BC | CVA | | Δ | BC | CVA | | Δ | BC | CVA | | Δ |
| | (letter | s read) | (letter | s read) | (letter | s read) | (letter | s read) | (letter | s read) | (letter | rs read) |
| | Study | Fellow | Study | Fellow | Study | Fellow | Study | Fellow | Study | Fellow | Study | Fellow |
| Visit | Eye | Eye | Eye | Eye | Eye | Eye | Eye | Eye | Eye | Eye | Eye | Eye |
| Baseline | • | - | • | | - | | • | | • | <u> </u> | • | |
| N | X | X | | | X | X | | | X | X | | |
| Median | X.X | X.X | | | X.X | X.X | | | X.X | X.X | | |
| Mean (SD) | x(x) | x (x) | | | x(x) | x (x) | | | x(x) | x(x) | | |
| (Min, Max) | (x, x) | $(\mathbf{x}, \mathbf{x})$ | | | (x, x) | $(\mathbf{x}, \mathbf{x})$ | | | (x, x) | $(\mathbf{x}, \mathbf{x})$ | | |
| Month 1 | | | | | | | | | | | | |
| N | X | X | X | X | X | X | X | X | X | X | X | X |
| Median | X.X | X.X | X.X | X.X | X.X | X.X | X.X | X.X | X.X | X.X | X.X | X.X |
| Mean (SD) | x(x) | x (x) | x(x) | x (x) | x(x) | x(x) | x (x) | x (x) | x(x) | x (x) | x (x) | x(x) |
| (Min, Max) | (x, x) | (x, x) | (x, x) | (x, x) | (x, x) | (x, x) | (x, x) | (x, x) | (x, x) | (x, x) | (x, x) | (x, x) |
| Change of $\geq 10$ letters, N(%) <sup>1</sup> | | x (x%) | | x (x%) | | x (x%) | | x (x%) | | x (x%) | | x (x%) |
| Month 2 | | | | | | | | | | | | |
| ••• | | | | | | | | | | | | |
| ••• | | | | | | | | | | | | |
| Month 24 | | | | | | | | | | | | |

 $\Delta$  indicates change from baseline.

<sup>&</sup>lt;sup>1</sup> Denominators are the number of participants in the safety population in each treatment arm and overall with data at the given visit. Percentages are rounded to the nearest whole number.

February 18, 2021

## **Table 18: Summary of Central Retinal Thickness Over Time**

This table will be similar to Table 17. The row corresponding to Change of  $\geq$  10 letters will be excluded.

## **Table 19: Summary of IOP Over Time**

This table will be similar to Table 17. The row corresponding to Change of  $\geq$  10 letters will be excluded.

Table 20: Results of Thyroid Palpation Assessment and Review of Systems Over Time

| | | Minoc | ycline | | | Plac | ebo | | | To | tal | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Significant<br>Findings | Re | view of Syste | ems | Significant<br>Findings | Re | view of Syste | ems | Significant<br>Findings | Re | view of Syste | ems |
| | Thyroid | | Sun | | Thyroid | | Sun | | Thyroid | | Sun | |
| Visit | <b>Palpation</b> | <b>Dizziness</b> | Sensitivity | Diarrhea | Palpation | <b>Dizziness</b> | Sensitivity | Diarrhea | Palpation | <b>Dizziness</b> | Sensitivity | Diarrhea |
| Baseline | - | | <u> </u> | | | | | | | | <u> </u> | |
| Yes | x (x%) | | | | x (x%) | | | | x (x%) | | | |
| No | x (x%) | | | | x (x%) | | | | x (x%) | | | |
| Month 1 | , , | | | | ` , | | | | . , | | | |
| Yes | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) |
| No | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) |
| Month 2 | | | | | | | | | | | | |
| Yes | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) |
| No | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) |
| | , , | | , , | | , , | , , | | | , , | , , | | |
| Month 24 | | | | | | | | | | | | |
| Yes | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) |
| No | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) | x (x%) |

Denominators are the number of participants in the safety population in each treatment arm and overall with data at the given visit. Percentages are rounded to the nearest whole number.

**Table 21: Summary of Laboratory Assessments Over Time** 

| | | Minocyc | line | | | Placebo | ) | | | Total | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Participants with Lab | Abnormal<br>Lab | A nv. A | Clinically<br>Significant | Participants with Lab | Abnormal<br>Lab | Any A | Clinically<br>Significant | Participants with Lab | Abnormal<br>Lab | A ny A | Clinically<br>Significant |
| Visit | Assessments<br>N <sup>1</sup> | Assessments<br>N (%) <sup>2</sup> | Any Δ<br>N (%) <sup>2</sup> | $\frac{\Delta}{N}$ (%) <sup>2</sup> | Assessments<br>N <sup>1</sup> | Assessments<br>N (%) <sup>2</sup> | Any Δ<br>N (%) <sup>2</sup> | $\frac{\Delta}{N}$ (%) <sup>2</sup> | Assessments<br>N <sup>1</sup> | Assessments<br>N (%) <sup>2</sup> | Any Δ<br>N (%) <sup>2</sup> | $N (\%)^2$ |
| Baseline | X | x (%) | 11 (70) | 1 ( / 0 ) | X | x (%) | 1 (70) | 1 (70) | X | x (%) | 11(70) | 11 (70) |
| Month 2 | X | . , | x (%) | x (%) | X | . , | x (%) | x (%) | X | ` ' | x (%) | x (%) |
| Month 6 | X | | x (%) | x (%) | X | | x (%) | x (%) | X | | x (%) | x (%) |
| Month 10 | X | | x (%) | x (%) | X | | x (%) | x (%) | X | | x (%) | x (%) |
| | X | | x (%) | x (%) | X | | x (%) | x (%) | X | | x (%) | x (%) |
| ••• | X | | x (%) | x (%) | X | | x (%) | x (%) | X | | x (%) | x (%) |
| Month 22 | X | | x (%) | x (%) | X | | x (%) | x (%) | X | | x (%) | x (%) |
| Month 24 | X | | x (%) | x (%) | X | | x (%) | x (%) | X | | x (%) | x (%) |

 $\Delta$  indicates changes from baseline

<sup>&</sup>lt;sup>1</sup> Participants in the safety population in each treatment arm and overall with laboratory assessment data at the given visit.
<sup>2</sup> Denominators are the number of participants in the safety population in each treatment arm and overall with laboratory assessment data at the given visit.

## **FIGURES**

Figure 1: Consort Diagram



Figure 2: Mean Best-Corrected Visual Acuity Over Time by Treatment Arm





Figure 3: Best-Corrected Visual Acuity Over Time by Participant

Figure 4: Mean Central Retinal Thickness Over Time by Treatment Arm This figure will be similar to Figure 2.

Figure 5: Central Retinal Thickness Over Time by Participant

This figure will be similar to Figure 3.

## **LISTINGS**

**Listing 1: Demographic Information by Participant** 

| Site | Participant<br>ID | Treatment<br>Arm | Registration<br>Date | Study<br>Eye | Age | Gender | Race | Ethnicity |
|---|---|---|---|---|---|---|---|---|
| XXX | 001 | XX | mm/dd/yy | XX | XX | XXX | XXX | XXX |
| XXX | 002 | XX | mm/dd/yy | XX | XX | XXX | XXX | XXX |
| | ••• | ••• | ••• | | | | | |

**Listing 2: IP Compliance** 

| Site | Participant<br>ID | Treatment<br>Arm | Number of<br>Doses Taken | Number of<br>Doses Missed | Expected Number of Doses Taken | Compliance<br>Rate (%) |
|---|---|---|---|---|---|---|
| XXX | 001 | XX | XX | XX | XX | X.X |
| XXX | 002 | XX | XX | XX | XX | X.X |
| | ••• | | ••• | | ••• | |

## **Appendix: Assessment of COVID-19 Impacts**

**Listing A1. Visit Schedule Deviations Due to COVID-19** 

| Participant ID | Visit Number | Type of Deviation |
|----------------|--------------|------------------------|
| 001 | Month X | Missed / Out-of-Window |
| | Month X | Missed/Out-of-Window |
| 002 | Month X | Missed/Out-of-Window |
| | Month X | Missed/Out-of-Window |
| | Month X | Missed/Out-of-Window |